CLINICAL TRIAL: NCT05352958
Title: Contribution of Diaphragmatic Ultrasound for Monitoring Diaphragmatic Function in Patients With Amyotrophic Lateral Sclerosis
Acronym: ALSUS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GEORGES 2021
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Amyotrophic Lateral Sclerosis: ALS
  * certain or probable according to the revised Escorial criteria
  * no indication for non-invasive ventilation
  Interventions: Procedure: Diaphragmatic ultrasound; Other: Electro-physiological exploration of the diaphragm

INTERVENTIONS:
Procedure: Diaphragmatic ultrasound — duration 15 minutes, performed at M0, M3, M6 and M9
Other: Electro-physiological exploration of the diaphragm — duration between 30 and 60 minutes performed at M0

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a rare neuromuscular disease that occurs in adults. It is characterized by a progressive degeneration of the first and second motor neurons leading to muscle failure. In its spinal form, ALS manifests by a progressive worsening of limb involvement, whereas the bulbar form presents with swallowing disorders, dysarthria and feeding difficulties.

Respiratory impairment is the most serious feature of ALS. Phrenic nerve damage causes diaphragmatic weakness, which inevitably leads to chronic restrictive respiratory failure. At the stage of symptomatic nocturnal or diurnal alveolar hypoventilation, non-invasive ventilation (NIV) prolongs survival while improving quality of life by relieving respiratory symptoms.

The indication for the initiation of NIV is based on the appearance of respiratory symptoms but also on the demonstration of diaphragmatic insufficiency. A quarterly follow-up of diaphragmatic function has been recommended by the French Health Authority since 2006. It is based on functional respiratory explorations (VC in sitting and lying position, measurement of maximal inspiratory pressure) and screening for diurnal or nocturnal hypoventilation with the measurement of PaCO2 or the nocturnal recording of SpO2.

Access to these examinations remains limited and they are sometimes complex to perform (in particular issues with mouth occlusion during respiratory manoeuvres in case of bulbar damage). Thus, only 60% of patients undergo a complete evaluation. Moreover, these explorations are only late markers of diaphragmatic dysfunction, and it has recently been shown that they do not correlate with histological diaphragmatic amyotrophy.

The development of new, reliable, and easily available tools for the evaluation of diaphragmatic function, and that are capable of detecting diaphragmatic insufficiency early in the course of the disease, are therefore necessary. Such tools would make it easier to implement NIV at the optimal time, preventing episodes of acute respiratory distress.

Recently, diaphragmatic ultrasound has appeared in the ICU as a new tool for assessing diaphragmatic function. It has the advantage of being highly available, inexpensive, non-irradiating, quick to perform, reproducible and very sensitive and specific for the diagnosis of diaphragmatic dysfunction.

In ALS, few studies have investigated the contribution of ultrasound for the diagnosis or follow-up of diaphragmatic dysfunction. In addition, no study so far has compared diaphragmatic ultrasound to complete pulmonary function test (PFT) data or to direct measurement of diaphragmatic pressure (Pdi). Very few publications report the how the diaphragm changes on ultrasound imaging during the disease. Moreover, these studies do not analyse the interest of diaphragmatic ultrasound in the prediction of progression towards respiratory failure with respiratory support, or death. Finally, these studies use different ultrasound measurements of the diaphragm (stroke, thickness, thickening fraction, and thickening fraction ratio, among others) rather than a simple, consensual parameter.

The aim of this study is to describe the evolution of diaphragmatic ultrasound parameters, to identify the parameter that best correlates with other respiratory measures (PFT, PaCO2, nocturnal oximetry) and to determine the prognostic value of diaphragmatic ultrasound in predicting the initiation of NIV or death at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Amyotrophic Lateral Sclerosis

  * Certain or probable according to the revised Escorial criteria
  * no indication for non-invasive ventilation
* Adult patient
* Patient who has given oral consent
* Patient who speaks and reads French

Exclusion Criteria:

* Patients with pre-existing diaphragmatic dysfunction requiring non-invasive ventilation
* Person who is not affiliated to national health insurance
* Person subject to a legal protection measure (curatorship, guardianship)
* Patients deprived of their liberty
* Pregnant, parturient or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Amyotrophic Lateral Sclerosis with no indication for non-invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Ultrasound measurement of the diaphragmatic stroke | Up to Month 9
Ultrasound measurement of diaphragmatic thickness | Up to Month 9

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No